CLINICAL TRIAL: NCT02033616
Title: Phase II, Double-Blind, Randomized Trial Of AVOVA-1 (Autologous Dendritic Cells Loaded With Autologous Tumor Associated Antigens) Vs. Autologous Peripheral Blood Mononuclear Cells (MC) In Patients With Stage III Or IV Epithelial Ovarian, Fallopian Tube Or Primary Peritoneal Carcinoma After Primary Therapy
Brief Title: Autologous Dendritic Cells Loaded With Autologous Tumor Associated Antigens for Treatment of Advanced Epithelial Ovarian Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aivita Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-OVA-P01
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Stage III Ovarian Carcinoma; Stage IV Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVOVA-1 (Experimental): Autologous dendritic cells loaded with tumor associated antigens (TAA) from autologous self-renewing tumor cells. AVOVA-1 is admixed with granulocyte-macrophage colony stimulating factor (GM-CSF) as an adjuvant, prior to injection.
  Interventions: Biological: AVOVA-1
- MC (Placebo Comparator): Autologous monocytes will serve as the control arm. MC is admixed with GM-CSF as an adjuvant, prior to injection.
  Interventions: Biological: MC

INTERVENTIONS:
Biological: AVOVA-1 — Comparison of a cancer treatment containing autologous dendritic cells loaded with tumor associated antigens (TAA) from autologous self-renewing tumor cells vs. a cancer treatment containing autologous immune cells.
  Arms: AVOVA-1
Biological: MC — Comparison of a cancer treatment containing autologous dendritic cells loaded with tumor associated antigens (TAA) from autologous self-renewing tumor cells vs. a cancer treatment containing autologous immune cells.
  Arms: MC

SUMMARY:
This is a double-blind study in which approximately 99 study patients will be randomized in a 2:1 ratio to receive either AVOVA-1 or MC. Patients eligible for randomization and treatment will be those (1) who have undergone debulking surgery, (2) for whom a cell line has been established, (3) who have undergone leukapheresis from which sufficient PMBC were obtained, and (4) have an ECOG performance grade of 0 or 1 (Karnofsky score of 70-100%).

The primary endpoint of this trial is death from any cause with the metric of OS from the date of randomization. PFS will be a secondary endpoint and will be calculated as the time from the date of randomization for treatment until subjective tumor progression or death. Progression will be subjectively defined by the treating physician, and is expected to be based on tumor marker levels (e.g. CA-125) and/or imaging. Secondarily, we will also define PFS and OS from the date of debulking surgery.

Patients will be stratified into (1) no evidence of disease (NED) (no measurable or non-measurable disease per RECIST and normal CA-125 levels) or (2) non-NED (measurable or non-measurable disease per RECIST or elevated CA-125 levels).

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-1 (Karnofsky score of 70-100%)
* Successful establishment of an autologous epithelial ovarian, fallopian tube, or primary peritoneal cancer cell line by AIVITA Biomedical, Inc.
* Patients must previously have been staged as having stage III [intraperitoneal (IP)] or Stage IV (distant metastatic) ovarian, fallopian tube, or primary peritoneal cancer, have undergone surgical debulking, and have initiated or completed standard adjuvant chemotherapy, which may include intravenous (IV) and/or IP chemotherapy using standard regimens. Patients will be characterized as being NED or non-NED per physical exam, CT and/or PET scans, and CA-125.
* Have undergone leukapheresis from which sufficient provided PBMC were obtained to produce an investigational treatment.
* Patients with one or a few brain metastases that have been treated with stereotactic radiotherapy consisting of a single dose, such as Gamma Knife or Cyberknife, are allowed to be included in the study, but need wait one week after such treatment.
* Written informed consent for treatment with investigational treatment

Exclusion Criteria:

* Known to have active hepatitis B or C or HIV
* ECOG performance status greater than 1 (Karnofsky score less than 70%).
* Known underlying cardiac disease associated with myocardial dysfunction that requires active medical treatment, or unstable angina related to atherosclerotic cardiovascular disease, or under treatment for arterial or venous peripheral vascular disease
* Diagnosis of any other invasive cancer or other disease process which is considered to be life-threatening within the next five years, and/or taking anti-cancer therapy for cancer other than ovarian (such as continuation of hormonal therapy for prostate or breast cancer diagnosed more than five years earlier).
* Active infection or other active medical condition that could be eminently life-threatening, including active blood clotting or bleeding diathesis.
* Active central nervous system metastases at the time of treatment.
* Known autoimmune disease, immunodeficiency, or disease process that involves the use of immunosuppressive therapy.
* Received another investigational drug within 28 days of the first dose or are planning to receive another investigational drug while receiving this investigational treatment.
* Known hypersensitivity to GM-CSF

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2017-11-18 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Overall Survival | 5 years
  Overall Survival: time to death from date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Aivita Biomedical, Inc.
Locations (6):
- United States (6):
  - Disney Family Cancer Center, Burbank, California
  - Scripps Health, La Jolla, California
  - UC San Diego, Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Irvine, Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Hospital - Cancer Center, Aurora, Colorado